CLINICAL TRIAL: NCT04032691
Title: The Effects of Alpha-2 Adrenergic Receptor Modulation on Rates of Carbon-11 Butanol Clearance From Ventricular Cerebrospinal Fluid
Brief Title: PET Study of a2a Agonist Effects on the Ventricular CSF Clearance of [11C]Butanol
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-05020048
Record Dates: First submitted 2019-07-19; First posted 2019-07-25 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Clonidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Clonidine Pill (Experimental): 0.1 mg by mouth daily at bedtime for one week
  Interventions: Drug: Clonidine Pill

INTERVENTIONS:
Drug: Clonidine Pill — 0.1 mg by mouth daily at bedtime for one week
  Other Names: On-Drug

SUMMARY:
This investigator initiated, pilot study will assess the feasibility of characterizing the effects of an orally administered alpha-2 adrenergic (a2a) agonist, clonidine, on the clearance rates of Carbon-11 butanol from the ventricular cerebrospinal fluid (vCSF) with positron emission tomography (PET) in healthy volunteers.

DETAILED DESCRIPTION:
This will be an open label pilot study of feasibility in healthy volunteers with no therapeutic intent. Vital signs, electrocardiogram (ECG) parameters, and sleep quality will be measured repeatedly during a one week lead-in period. Then, the ventricular cerebrospinal fluid (vCSF) clearance rates of [11C]butanol will be measured with PET before and after one week of treatment with clonidine, 0.1 mg by mouth daily at bedtime. Safety surveillance will be augmented with home health monitoring devices that are wifi and blue tooth enabled. Surveillance for adverse events related to drug discontinuation will be monitored for one week during a washout period.

Primary Objective: To assess the logistical feasibility and safety of treating normotensive adults with clonidine and monitoring its effects with home health devices. The primary outcome measure will be the number of adverse events (AEs) or serious adverse events (SAEs). Other measures will include changes in sleep quality, vital signs and ECG parameters, such as the PR and corrected QT intervals.

Secondary Objectives: To estimate drug-induced changes in vCSF clearance rates of butanol with PET scans acquired before and after treatment as a function of steady-state plasma levels of clonidine.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent. No vulnerable populations.
* Age 18-to-89 years old
* Mini-Mental Status Examination of ≥ 28
* Confirmed by the screening procedures to still be reasonably healthy and, in the opinion of the investigators, likely to tolerate the imaging procedures. For example, patients with chronic low back pain might not be able to lie still for very long.
* Confirmed by the screening procedures to have normal hemodynamic function. Systolic blood pressure and pulse must be higher than 120 mmHg and 60 beats per minute (bpm) while sitting. At the discretion of the investigators, athletic people who engage in vigorous exercise of one hour or more at least four times per week may be enrolled if their systolic blood pressure and pulse are higher than 100 mmHg and 50 beats per minute while sitting.
* Unremarkable electrocardiograms with PR intervals of less than 200 mSec and QT interval corrected with Frederica's method (QTcF) of less than 440 mSec.
* Willing and able to refrain from abusing any recreational drugs, including marijuana because of its sleep effects, and drink less than one unit of alcoholic beverages per day starting one week prior to the lead-in period, and avoided for the next three weeks while on study (the one week lead-in period, one week on drug period, and one week washout period).
* Willing to refrain from donating blood during the month of study (because of its potential effect of quickening pulse).
* Willing to refrain from participating in any other research study that requires taking medication during the month of study.
* Willing to refrain from being vaccinated during the month of study.
* Have not participated in research with exposure to ionizing radiation that would result in approaching the exposure limits for healthy volunteers described in the Code of Federal Regulations, Title 21 Part 361.1 (21CFR361.1)

Exclusion Criteria:

* History of allergy to clonidine.
* History of multiple hypersensitivity reactions, as indicated by allergies to multiple medications, foods, and seasonal pollens.
* History or physical examination suggestive of a condition, disorder, or disease that could represent a contra-indication to taking an antihypertensive. The relative contraindications to clonidine listed in the package insert under the section on precautions will be exclusionary in this study. They include subjects with coronary artery insufficiency syndromes, histories of myocardial infarction, cardiac conduction abnormalities, cerebrovascular disease, and chronic renal failure.
* Women who are pregnant or breast feeding will not be eligible to participate in the study, as clonidine is classified as a Class C risk to a fetus. (In fact, there is a safety signal in pregnant animal models that justifies exclusion, even if the signal is weak.)
* History, physical examination or clinical laboratory test result suggestive of a condition, disorder, or disease that could affect the adsorption, distribution, metabolism or excretion of clonidine, including an alcohol abuse or dependence disorder.
* Positive urine toxicology screen for drugs other than cannabis.
* Subjects may not be a member of a vulnerable population.
* May not have donated blood in the 30 days prior to the start of the lead-in period.
* May not have participated in research administering drugs in the last 30 days.
* May not have been vaccinated in the 30 days prior to the start of the lead-in period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-05-24 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | one week on drug
  Clinically significant changes in hemodynamic function, including vital signs (VSs) and ECG parameters, will be classified as adverse events.

SECONDARY OUTCOMES:
Change in Ventricular CSF Clearance Rates of [11C]Butanol | after one week on drug compared to drug free baseline rates
  The rate of change in the concentration of radioactivity as a function of time before drug treatment compared to after drug treatment.

OTHER OUTCOMES:
Sleep Quality: Duration | Average of one week before drug compared to one week on drug, and one week after drug.
  Time interval between falling asleep and waking up as estimated with a wearable sleep tracker.
Sleep Quality: Time in Deep Sleep | Average of one week before drug compared to one week on drug, and one week after drug.
  Sum of time intervals classified as representing deep sleep by a wearable sleep tracker.
Sleep Quality: number of nocturnal awakenings | Average of one week before drug compared to one week on drug, and one week after drug.
  Number of times that nocturnal activity is classified as an awakening by a wearable sleep tracker.
Sleep Quality: Subjective Self Rating of Quality | Component and global scale scores on Day 1 (before drug) compared to score on Day 2 (after first dose of drug), Day 8 (after one week on drug) and Day 16 (after one week of washout).
  Score on each component and the "global" sum of subscale scores on the Pittsburgh Sleep Quality Index (PSQI), where the range of scores on the seven components varies from 0 (good sleep) through 3 (bad sleep).

CONTACTS AND LOCATIONS:
Overall Officials: P. David Mozley, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The safety data will be shared. Data will be from the lead-in period, the on-drug period, and the washout period. Safety data include vital signs, electrocardiogram parameters, and quality of sleep measures.
Supporting Information: Study Protocol, CSR
Time Frame: Available at end of study (anticipated date = 31 Dec 2020) for up to five years.
Access Criteria: All investigators who provide a brief statement expressing a scientific interest.